CLINICAL TRIAL: NCT00352430
Title: Cardiopulmonary Function Assessment and NO Based Therapies for Patients With Hemolysis-Associated Pulmonary Hypertension
Brief Title: Cardiopulmonary Function Assessment and NO-Based Therapies for Patients With Hemolysis-Associated Pulmonary Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060202; 06-H-0202
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2015-12-07

CONDITIONS: Pulmonary Hypertension
Keywords: Nitric Oxide; PDE Inhibitors; Pulmonary Hypertension; Sickle Cell; Thalassemia; Sickle Cell Anemia
MeSH Terms: conditions — Hypertension, Pulmonary; Thalassemia; Anemia, Sickle Cell

INTERVENTIONS:
Drug: Nitric Oxide/INP Pulse Delivery
Drug: Nitric Oxide/INO Pulse Delivery

SUMMARY:
This study will evaluate new treatments for people who have pulmonary hypertension, or high blood pressure in the lungs, caused by sickle cell anemia or thalassemia.

Patients ages 18 and older with a diagnosis of sickle cell disease or thalassemia, who have mild to severe pulmonary hypertension, and who are not pregnant or breastfeeding may be eligible for this study. There are three stages in the study, with up to 200 participants in the screening. Patients will undergo pulmonary function tests, including those for asthma and measurement of oxygen levels in the arterial blood. They will have a chest X-ray, computed tomography (CT) scan of the lungs, ventilation perfusion lung scan to look for blood clots, echocardiogram, test to measure how far patients can walk in 6 minutes, nighttime oxygen measurement done while asleep, blood collection, magnetic resonance imaging (MRI) scan of the heart, and exercise test. About 3 to 4 days are needed for the tests, all of which can be done while patients are outpatients, except for the sleep study. For the CT scan, patients lie on a table while an X-ray beam takes images of the lungs and heart. The lung scan involves breathing of a small amount of a radioactive aerosol called Tc99m DTPA while pictures are taken of the lungs from various angles. Then an injection of albumin, a protein with a small amount of radioactivity, will be given, and more lung pictures will be taken. For the MRI scan, patients lie on a table that slides into a machine. A medication called gadolinium will be injected, to help improve images made through the scan. After the tests, patients will be admitted to the Clinical Center for 1 day. A small plastic catheter, or tube, will be placed in the vein of an arm. A longer catheter will go into a deeper vein (neck or leg), and a pulmonary artery catheter will be inserted to measure blood pressure in the blood vessels. Doctors will guide the catheter into the lung artery. Patients will be asked to pedal on a stationary bicycle while heart and lung pressure is measured. If pulmonary hypertension is present, patients will proceed to the second stage (up to 50 participants). While the catheter is still in place, patients will wear a face mask and breathe nitric oxide (NO) for 20 minutes. They will take 50 mg of sildenafil by mouth, and pressure in the heart and lungs will be monitored for about 4 hours. They will again receive NO for another 20 minutes. Blood samples will be taken, and the heart rhythm and pressure in the lungs will be monitored. Sildenafil can cause headache, flushing, and indigestion. Side effects of the lung scan involve allergic reactions to DTPA and albumin. Patients with an allergy to eggs should not have that test.

Up to 25 patients can enter the third stage. They will breathe NO by using a tank of gas that delivers it through tubes to the nose, for a period of 6 weeks. They will continue taking sildenafil as previously prescribed and visit the clinic every 2 to 4 weeks for an echocardiogram, blood tests, and 6-minute walk test. After 6 weeks, patients will have catheterization of the heart again to measure pressure in the heart and lungs. Then NO will be stopped, and pressure in the lungs will be checked to see if NO has helped lower the blood pressure-and to make sure that the blood pressure does not increase when medication is stopped. Patients whose symptoms have improved as a result of breathing NO may wish to continue with that therapy.

DETAILED DESCRIPTION:
Sickle cell anemia is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Acute pain crisis, acute chest syndrome (ACS), and secondary pulmonary hypertension are common complications of sickle cell anemia. Pulmonary hypertension has now been identified as a major cause of death in adults with sickle cell disease. Similarly, pulmonary hypertension has been identified as a chronic complication of hemolytic disorders such as thalassemia, hereditary spherocytosis and paroxysmal nocturnal hemoglobinuria. Sildenafil has been proposed as a possible therapy for both primary and secondary pulmonary hypertension and recent phase I/II studies from the intramural NIH suggest it is well tolerated and efficacious in this population. Furthermore, a number of recent studies have suggested that NO based therapies may have a favorable impact on sickle red cells at the molecular level and could improve the abnormal microvascular perfusion that is characteristic of sickle cell anemia.

This clinical trial is designed with three major objectives: 1) to assess cardiopulmonary function in patients with sickle cell disease and thalassemia with and without pulmonary hypertension, 2) to determine the relative acute vasodilatory effects of sildenafil, and inhaled NO in patients with hemolysis-associated pulmonary hypertension and 3) to determine the chronic effects of the addition of inhaled NO on pulmonary hemodynamics and functional capacity in patients with hemolysis-associated pulmonary hypertension chronically treated with sildenafil.

ELIGIBILITY:
* INCLUSION CRITERIA
* Males or females, 18 years of age or older.
* Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or S thalassemia genotype is required) or thalassemia.
* For female subjects, on a reliable method of birth control or not physically able to bear children.

<TAB>

For Stage II:

* Mild to severe pulmonary hypertension with mean pulmonary artery pressure greater than 25 mm Hg at rest or greater than 30 mm Hg during exercise, measured by pulmonary artery catheterization.
* Pulmonary artery wedge pressure or left ventricular end-diastolic pressure less than or equal to 18 mm Hg or gradient between pulmonary artery diastolic pressure and wedge pressure greater than 8 mm Hg or echocardiographic criteria to exclude left ventricular dysfunction.
* For female subjects, on a reliable method of birth control or not physically able to bear children.

For Stage III:

* Mild to severe pulmonary hypertension with mean pulmonary artery pressure greater than 25 mm Hg at rest or greater than 30 mm Hg during exercise, measured by pulmonary artery catheterization in patients on chronic sildenafil therapy for at least three months. Patients receiving combination drug therapy with other drugs (e.g., endothelin antagonists, prostacyclins) are allowed to participate in stage III as long as sildenafil is one of the components of the combination regimen.
* Pulmonary artery wedge pressure or left ventricular end-diastolic pressure less than or equal to 18 mm Hg or gradient between pulmonary artery diastolic pressure and wedge pressure greater than 8 mm Hg or echocardiographic criteria to exclude left ventricular dysfunction.
* Must be on chronic sildenafil therapy on a stable dose for at least three months.
* For female subjects, on a reliable method of birth control or not physically able to bear children.

EXCLUSION CRITERIA

For Stage I

* Current pregnancy or lactation.
* Any condition that in the opinion of the study investigators would adversely affect the outcome of the study or the safety of the volunteer.

For Stage II and III:

* Current pregnancy or lactation.
* Any of the following medical conditions

  1. Stroke within the last six weeks.
  2. History of sustained priapism requiring medical or surgical treatment, unless currently impotent or on exchange transfusion therapy, within two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-07-09; Primary Completion 2010-03-10 (Actual); Study Completion 2010-03-10 (Actual)

PRIMARY OUTCOMES:
To assess cardiopulmonary function in patients with sickle cell disease and thalassemia with and without pulmonary hypertension.

SECONDARY OUTCOMES:
To determine the relative acute vasodilatory effects of sildenafil, and inhaled NO in patients with hemolysis-associated pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Castro O. Systemic fat embolism and pulmonary hypertension in sickle cell disease. Hematol Oncol Clin North Am. 1996 Dec;10(6):1289-303. doi: 10.1016/s0889-8588(05)70401-9. PMID 8956017
- [Background] Sutton LL, Castro O, Cross DJ, Spencer JE, Lewis JF. Pulmonary hypertension in sickle cell disease. Am J Cardiol. 1994 Sep 15;74(6):626-8. doi: 10.1016/0002-9149(94)90760-9. No abstract available. PMID 8074054
- [Background] Norris SL, Johnson C, Haywood LJ. Left ventricular filling pressure in sickle cell anemia. J Assoc Acad Minor Phys. 1992;3(1):20-3. PMID 1576456
- [Derived] Nguyen KL, Tian X, Alam S, Mehari A, Leung SW, Seamon C, Allen D, Minniti CP, Sachdev V, Arai AE, Kato GJ. Elevated transpulmonary gradient and cardiac magnetic resonance-derived right ventricular remodeling predict poor outcomes in sickle cell disease. Haematologica. 2016 Feb;101(2):e40-3. doi: 10.3324/haematol.2015.125229. Epub 2015 Nov 20. No abstract available. PMID 26589907
- [Derived] Wang X, Mendelsohn L, Rogers H, Leitman S, Raghavachari N, Yang Y, Yau YY, Tallack M, Perkins A, Taylor JG 6th, Noguchi CT, Kato GJ. Heme-bound iron activates placenta growth factor in erythroid cells via erythroid Kruppel-like factor. Blood. 2014 Aug 7;124(6):946-54. doi: 10.1182/blood-2013-11-539718. Epub 2014 Jun 10. PMID 24916507
- [Derived] Villagra J, Shiva S, Hunter LA, Machado RF, Gladwin MT, Kato GJ. Platelet activation in patients with sickle disease, hemolysis-associated pulmonary hypertension, and nitric oxide scavenging by cell-free hemoglobin. Blood. 2007 Sep 15;110(6):2166-72. doi: 10.1182/blood-2006-12-061697. Epub 2007 May 29. PMID 17536019